CLINICAL TRIAL: NCT01104051
Title: A Prospective, Single Center, Double Blind, Randomized, Sham Controlled, Crossover Study to Evaluate the Clinical Efficacy of Radiofrequency Nerve Ablation Using Simplicity III Versus Sham for the Treatment of Chronic Low Back Pain Associated With Sacroiliac Joint Dysfunction
Brief Title: Radiofrequency Nerve Ablation Versus Sham to Treat Chronic Low Back Pain Caused by Sacroiliac Joint Dysfunction
Status: Completed | Type: Observational
Sponsor: Coastal Orthopedics & Sports Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: RBSI001
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Sacroiliac Joint Dysfunction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Radiofrequency Ablation: The treatment to be used in this trial is radiofrequency nerve ablation of lateral branches from S1 - S4 using radiofrequency treatments; Simplicity lll Electrode, a single RF electrode with a single percutaneous entry point.
- Sham: subjects to be blinded,to receive sham procedure; The treatment to be used in this trial is radiofrequency nerve ablation of lateral branches from S1 - S4 using radiofrequency treatments; Simplicity lll Electrode, a single RF electrode with a single percutaneous entry point.

SUMMARY:
Trial will enroll qualified subjects at a 2:1 ration to receive radiofrequency ablation or sham. At six weeks follow up they will be unblinded; sham subjects will then be given option to receive treatment.

Subjects will be followed after procedure for data collection for economic outcomes and efficacy of treatment.

DETAILED DESCRIPTION:
Patients presenting with low back pain associated with SIJD for longer than 6 months, and who have not had positive responsive to the conservative treatments:

* Pharmacologic Management
* Therapies; physical, acupuncture, massage etc…
* Other alternative treatments

Enrollment, Treatment/Sham Procedure, Follow-up at 3 weeks, 6 weeks with unblinding, 4, 6, 9 months. Un-blinding occurring at 6 weeks with crossover option to receive treatment. Total visits 7 with enrollment approximately over a period of 9 months. Trial extension optional for phone contact at year 1, 2. Sham subjects receiving treatment will be followed at months 6 weeks, 4, and 6 months with phone calls at year 1, 2.

Patients who complete at least 50% of their patient diaries, and miss no more 2 consecutive office visits. Data will be used if patients have remained enrolled thru 4 month visit.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 years old, or older 2. Unilateral or Bilateral LBP or Buttocks Pain for greater than six months with a 3 day average VAS greater or equal to 4 on a 1-10 scale 3. Tenderness over the SI joint 4. 75% or greater relief of pain (with return to baseline) during the local anesthetic phase of two separate, one fluoroscopically guided intra-articular SI joint injection and one lateral branch block (see Appendix A) 5. Stable medications for pain for the last seven days 6. Have used at least 3 alternative treatments for pain without success (se 7. BMI less than 35.0

Exclusion Criteria:

1. Focal Neurologic Signs
2. Any component of pain related to Lumbar Z-joints at L4-5 and/or L5-S1 as determined by one set of medial branch blocks
3. Previous radiofrequency procedure within the last 6 months
4. Moderate or greater spinal stenosis
5. Greater than Grade 2 listhesis
6. Foraminal Stenosis; marked to severe
7. Previous Lumbar Spine Surgery
8. Unstable Medical or Psychological Conditions as determined by the investigator
9. Concomitant cervical or thoracic pain greater than 2/10 on VAS
10. Workers compensation, disability or litigation
11. Pregnancy, breast feeding or planning on becoming pregnant during the trial
12. Subject unwillingness to complete study related activities
13. Current Smoker; unless quit greater than 6 months -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with low back pain associated with SIJD for longer than 6 months, and who have not had positive responsive to the conservative treatments:
  * Pharmacologic Management
  * Therapies; physical, acupuncture, massage etc…
  * Other alternative treatments
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2010-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Reduction in pain | 6 months
  • To evaluate the clinical efficacy of RF lesioning of sensory innervation of the sacroiliac region as a long term treatment for pain associated with SI joint dysfunction as measured by the reduction in VAS scale and the use of pain alleviating therapies

SECONDARY OUTCOMES:
Economic outcomes | 1 year
  • To evaluate the economic and cost benefits of radiofrequency as a treatment for chronic pain associated with SI joint pain.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bundschu, MD, Principal Investigator — Coastal Orthopedics
Locations (1):
- Coastal Orthopedics & Sports Medicine, Bradenton, Florida, United States